CLINICAL TRIAL: NCT03599011
Title: Gustatory Dysfunction Among a Sample of Depressed Egyptian Adults Under Anti-depressants Therapy A Retrospective Cohort Study
Brief Title: Gustatory Dysfunction Among a Sample of Depressed Egyptian Adults Under Anti-depressants Therapy
Status: Completed | Type: Observational
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Christine Raouf George Mikhail, Principal Investigator, Cairo University
Other Study IDs: CEBD-CU-2018-07-21
Record Dates: First submitted 2018-07-16; First posted 2018-07-26 (Actual); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Taste Disorders
MeSH Terms: conditions — Taste Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Exposure 1: commonly prescribed tricyclic antidepressants (Imipramine, Amitriptyline, Clomipramine HCL) administered for at least 3 months
- Exposure 2: commonly prescribed Selective Serotonin Re-uptake inhibitors antidepressants ( Fluoxetine, Fluvoxamine, Sertraline, Citalopram, Paroxetine) administered for at least 3 months
- Non exposure: Non-pharmacological treatment (psychotherapy)

SUMMARY:
- Assess gustatory thresholds among a sample of depressed Egyptian adults (age from 20 to 50 years old) under anti-depressants therapy ( for at least 3 months) using filter paper disc(FPD) method through a scoring system. - Determine the taste intensity at supra-threshold among these patients using a psychophysical method through a scoring system. - Identify possible modulators for developing gustatory dysfunction among these patients using a questionnaire ( appendix) with a binary measuring unit (yes/no).

DETAILED DESCRIPTION:
PECO

* P Population: depressed Egyptian adults under anti-depressants therapy
* E1 Exposure 1: commonly prescribed tricyclic antidepressants (Imipramine, Amitriptyline, Clomipramine HCL)
* E2 Exposure 2: commonly prescribed Selective Serotonin Re-uptake inhibitors antidepressants ( Fluoxetine, Fluvoxamine, Sertraline, Citalopram, Paroxetine)
* C control (non exposure) : non-pharmacological treatment ( psychotherapy)
* O Outcome:

Primary 1ry : Assess gustatory thresholds among a sample of depressed Egyptian adults (age from 20 to 50 years old) under anti-depressants therapy ( for at least 3 months) using filter paper disc(FPD) method through a scoring system.

Secondary 2ry: - Determine the taste intensity at supra-threshold among these patients using a psychophysical method through a scoring system. - Identify gustatory dysfunction modulators among these patients using a questionnaire ( appendix) with a binary measuring unit (yes/no).

ELIGIBILITY:
Inclusion Criteria:

* Depressed Egyptian adults under antidepressants therapy for at least 3 months/non-pharmacological treatment( psychotherapy)
* Age from 20 to 50 years old

Exclusion Criteria:

* Antipsychotics
* Hypnotics
* Anticonvulsants
* Ages other than the mentioned
* Olfactory dysfunction
* Chemosensory dysfunction

Ages: 20 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: Depressed Egyptian adults under anti-depressants therapy The patients will be recalled using their phone numbers recorded in their follow up records in order to come to the Diagnosis center at the faculty of Dentistry, Cairo University to be assessed for gustatory functions and will be given identification numbers and divided into three groups, to which the operator shall be blinded.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2020-02-22 (Actual); Primary Completion 2020-08-08 (Actual); Study Completion 2020-10-07 (Actual)

PRIMARY OUTCOMES:
Gustatory thresholds | during anticipated period of 7 months from February 2020 till August 2020
  - C.M will assess the gustatory thresholds using filter paper disc method in which five concentrations of the substances will be used to test the four tastes: sweet, salty, sour and bitter and the concentrations of each taste shall be scored from disc number 1 (lowest) to number 5 (highest). - If the subject cannot detect the taste at the highest concentration, a score of 6 will be given. - The mean of three measurements for each test will be calculated.

SECONDARY OUTCOMES:
Taste intensity at supra-threshold | during anticipated period of 7months from February 2020 till August 2020
  - C.M will assess the taste intensity at supra-threshold level on a 9 point vertical labeled scale (extremely strong, very strong, strong, slightly strong, neutral, slightly weak, weak , very weak, extremely weak) in which subjects indicate the intensity perceived when tasting a substance
Gustatory dysfunction modulators | during anticipated period of 7months from February 2020 till August 2020
  -C.M will use an assessment questionnaire (appendix) to assess possible modulators for developing gustatory dysfunction including a number of short-term and long-term factors such as body mass, gender, age, local and systemic diseases, excessive alcohol drinking, drug dependence, smoking, state of oral hygiene, consumption of some foods or drugs

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Dentistry, Cairo University, Cairo, Egypt

REFERENCES:
- [Derived] Mikhail C, Elgaaly K, Abd El Latif Abd El Hamid A, Shaker O, Ali S. Gustatory Dysfunction among a Sample of Depressed Egyptian Adults under Antidepressants Therapy: A Retrospective Cohort Study. Int J Dent. 2021 Mar 4;2021:5543840. doi: 10.1155/2021/5543840. eCollection 2021. PMID 33747081